CLINICAL TRIAL: NCT00355758
Title: Prostate Cancer Detection by Serum Proteomic Profiling
Brief Title: UCI 03-72 Prostate Cancer Detection by Serum Proteomic Profiling
Status: Terminated | Type: Observational
Why Stopped: Lack of personnel
Sponsor: University of California, Irvine (Other)
Responsible Party: Atreya Dash, MD, University of California, Irvine
Other Study IDs: 2004-3561
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2010-09-01 (Estimated); Status verified 2010-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer Detection by Serum Proteomic Profiling
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood is collected from subjects. The whole blood is spun down by centrifugation and only serum is retained and stored.
Oversight: Data Monitoring Committee: No

SUMMARY:
: Researchers would like to see if a new test called SELDI (Surface Enhanced Laser Desorption Ionization) analysis can predict biopsy results better than PSA tests.

DETAILED DESCRIPTION:
A blood sample of approximately 30 cc will be collected prior to the patients standard of care radical prostatectomy surgery. This blood will be used for the SELDI analysis. The remainder of the blood sample will be stored and may be used for the PSA test at a later date. The patient will have a final blood draw 3 months to 1 year following surgery.

ELIGIBILITY:
Inclusion Criteria:

* For all subjects:

  * Men 50 years of age or older.
  * Serum PSA greater than or equal to 2.5 ng/ml and less then or equal to 10.0 ng/ml determined by a measurement within the past six months, and/or digital rectal exam suspicious for prostate cancer as determined by the patient's Urologist.
  * It has been determined by the treating physician that a prostate biopsy is clinically indicated.
  * Patients will have already been diagnosed with prostate cancer and scheduled for a radical prostatectomy.

For study on treatment effect

* Men with clinically localized prostate cancer (total PSA < 20 ng/ml and clinical T2b or less).
* Men with organ confined prostate cancer as determined by final pathologic diagnosis.

Exclusion Criteria:

* Exclusion criteria for all subjects:

  * Known prostate cancer or prior treatment for prostate cancer.
  * Acute prostatitis.
  * Untreated urinary tract infection.
  * Presence of Foley catheter or any urethral instrumentation in the previous 48 hours.
  * Hormonal therapies including LHRH agonists, oral anti-androgens, estrogenic compounds, Proscar or any phytotherapies within the previous 6 months.

Exclusion Criteria (for study on treatment effect)

* Men with non-organ confined prostate cancer.
* Men with detectable serum PSA levels more than 1 months following radical prostatectomy.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those who have prostate cancer and are scheduled for robotic prostatectomy to treat the disease and are seen at the Urology Clinic of the University of California, Irvine.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2005-04; Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atreaya Dash, MD, Principal Investigator — University of California
Locations (1):
- University of California, Irvine, Orange, California, United States